CLINICAL TRIAL: NCT05889312
Title: Improving Response Assessment in Cancer by Measurement of Cellular Redox Status Using 18F-FSPG Positron Emission Tomography
Brief Title: Assessing Cancer Treatment Response to Therapy Using 18F-FSPG PET
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 312860
Record Dates: First submitted 2023-05-16; First posted 2023-06-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Diagnosis; Resistant Cancer; Response, Acute Phase
MeSH Terms: conditions — Neoplasms; Disease; Acute-Phase Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-small cell lung cancer: NSCLC
  Interventions: Diagnostic Test: 18F-FSPG PET/CT in NSCLC
- Head and neck squamous cell cancer: HNSCC
  Interventions: Diagnostic Test: 18F-FSPG PET/CT in HNSCC

INTERVENTIONS:
Diagnostic Test: 18F-FSPG PET/CT in NSCLC — Stage 3 NSCLC with radical curative intent at baseline (pre-treatment) and at 4-8 weeks into treatment.
  Groups: Non-small cell lung cancer
Diagnostic Test: 18F-FSPG PET/CT in HNSCC — Stage 3 and 4 HNSCC with radical curative intent at baseline and at 2-4 weeks into treatment.
  Groups: Head and neck squamous cell cancer

SUMMARY:
Prospective single centre non-randomised exploratory observational study to measure changes in tumour cellular redox status with 18F-FSPG PET in stage 3 non-small cell lung cancer (NSCLC) and stage 3 and 4 head and neck squamous cell cancer (HNSCC) at baseline and during standard of care treatment, and to compare this with 18F-FDG PET/CT and RECIST 1.1 response at 12 weeks.

DETAILED DESCRIPTION:
Study design: Prospective single centre non-randomised exploratory observational study.

Number of patients: 32 (16 head and neck cancer, 16 lung cancer).

Primary hypothesis: Changes in 18F-FSPG uptake predict treatment efficacy.

Primary objectives: To measure changes in tumour cellular redox status with 18F-FSPG PET in stage 3 non-small cell lung cancer (NSCLC) and stage 3 and 4 head and neck squamous cell cancer (HNSCC) at baseline and during standard of care treatment, and to compare this with 18F-FDG PET/CT and RECIST 1.1 response at 12 weeks.

Secondary objectives: Characterise the uptake and pharmacokinetics of 18F-FSPG in NSCLC and HNSCC patients.

Determine the baseline level and variability of 18F-FSPG uptake within and between patients with NSCLC and HNSCC pre and post treatment.

Compare 18F-FSPG PET/CT imaging with standard measures of response (RECIST/PERCIST) and other clinical biomarkers (IHC and blood glutamate) at baseline and during cancer treatment.

Primary outcomes: Report and compare % change in 18F-FSPG uptake in NSCLC and HNSCC patients on standard of care treatment with standard measures of response (RECIST/PERCIST) Secondary outcomes: Report variation in 18F-FSPG uptake in NSCLC and HNSCC. Report kinetic data in 18F-FSPG uptake in NSCLC and HNSCC. Report correlation of 18F-FSPG uptake in NSCLC and HNSCC with available histology and blood markers.

Inclusion criteria:

1. Written informed consent
2. Aged 16 or above (as per NCRI)
3. Histologically confirmed NSCLC and HNSCC, who are treatment naïve and scheduled to commence standard of care treatment ((chemo)radiotherapy)
4. Willingness and ability to comply with scheduled study visits and tests
5. Confirmation of adequate function of all major organs and systems

Exclusion criteria :

1. Pregnant or lactating women
2. Concomitant uncontrolled medical conditions
3. Participants likely to require palliative radiotherapy within the first 12 weeks of treatment
4. Prognosis less than 3 months
5. Previous anti-cancer treatment (only treatment naïve patients eligible for inclusion)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged 16 or above
3. Histologically confirmed HNSCC or NSCLC, who are treatment naïve and scheduled to commence standard of care treatment ((chemo)radiotherapy)
4. Willingness and ability to comply with scheduled study visits and tests
5. Confirmation of adequate function of all major organs and systems

Exclusion Criteria:

1. Pregnant or lactating women
2. Concomitant uncontrolled medical conditions
3. Participants likely to require palliative radiotherapy within the first 12 weeks of treatment
4. Prognosis less than 3 months
5. Previous anti-cancer treatment (only treatment naïve patients eligible for inclusion)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: stage 3 non-small cell lung cancer (NSCLC) stage 3 and 4 head and neck squamous cell cancer (HNSCC)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Changes in tumour cellular redox status | 3 years
  To measure changes in tumour cellular redox status with 18F-FSPG PET in stage 3 non-small cell lung cancer (NSCLC) and stage 3 and 4 head and neck squamous cell cancer (HNSCC) at baseline and during standard of care treatment, and to compare this with 18F-FDG PET/CT and RECIST 1.1 response at 12 weeks.

SECONDARY OUTCOMES:
18F-FSPG kinetics | 2 years
  1. Characterise the uptake and pharmacokinetics of 18F-FSPG in NSCLC and HNSCC by measurement of tumour and normal tissue time activity curves time to peak
18F-FSPG heterogeneity | 3 years
  2. Determine the baseline level and variability of 18F-FSPG uptake within and between patients with NSCLC and HNSCC pre and post treatment
Correlation with histopathology and blood biomarkers | 3 years
  3. Correlation between 18F-FSPG PET/CT imaging standard measures of response (RECIST/PERCIST percent change) and percent change in other biomarkers (immunohistochemistry score and blood glutamate concentration) at baseline and during cancer treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only anonymised data will be shared.